CLINICAL TRIAL: NCT05485519
Title: Prospective, Randomized, Open Label Controlled Trial To Evaluate The Safety And Efficacy Of Dexmedetomidine Use Beyond 24 Hours Compared With Midazolam In Children Admitted To Pediatric Intensive Care Unit (PICU) at KASCH-MNGHA.
Brief Title: Prospective, Randomized, Open Label Controlled Trial To Evaluate The Safety And Efficacy Of Dexmedetomidine Use Beyond 24 Hours Compared With Midazolam In Children Admitted To Pediatric Intensive Care Unit at King Abdullah Specialist Children Hospital- Ministry of National Guard Health Affairs.
Acronym: PROMISE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC20/160/R
Record Dates: First submitted 2022-06-30; First posted 2022-08-03 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Dexmedetomidine; Midazolam; Withdrawal Symptoms; Failure of Extubation
Keywords: Dexmedetomidine; Midazolam; Intubation; Withdrawal Symptoms; failure of Extubating
MeSH Terms: conditions — Substance Withdrawal Syndrome | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (D) (Experimental): Infusion start at 0.5 mcg/kg/hour. Titrate to effect (up to1.5 mcg/kg/hour)
  Interventions: Drug: Dexmedetomidine
- Midazolam (M) (Active Comparator): 1 mcg/kg/minute. Up to a maximum of 5 mcg/kg/minute.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — Infusion start at 0.5 mcg/kg/hour. Titrate to effect (up to1.5 mcg/kg/hour)
  Arms: Dexmedetomidine (D)
Drug: Midazolam — (1 mcg/kg/minute. up to a maximum of 5 mcg/kg/minute.
  Arms: Midazolam (M)

SUMMARY:
Study will be conducted in Pediatric Intensive Care Unit (PICU) in King Abdullah Specialist Children Hospital (KASCH), National Guard Health Affairs, Riyadh, Saudi Arabia. Total of 430 patients will participate to assess the safety and efficacy of prolonged Dexmedetomidine use beyond 24 hours in pediatric Intensive Care Unite.

DETAILED DESCRIPTION:
Prospective, randomized, open label, controlled study, will be conducted in Pediatric Intensive Care Unit (PICU) in King Abdullah Specialist Children Hospital (KASCH), National Guard Health Affairs, Riyadh, Saudi Arabia. 340 patients will be randomly randomized to Midazolam (M) or Dexmedetomidine (D), to assess the safety and efficacy of prolonged Dexmedetomidine use beyond 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1-14 years both male and female who require mechanical ventilation
2. Informed consent from signed by patient's legal representatives, and for patients aged 12- 14 who has an age-appropriate understanding additional assent form signed by patient is required.
3. Intubated within 6 hours and anticipated to require mechanical ventilation for more than 48 hours

Exclusion Criteria:

1. Septic shock and/or multi-organ failure.
2. Hemodynamically instability and requires inotropes.
3. Severe intracranial or spinal trauma with high intracranial pressure
4. Liver failure
5. Acute or chronic renal failure.
6. Glasgow Coma Scale (GCS) ≤8
7. Known to have allergy to the study drugs
8. Airway surgery

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 430 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Mean time taken from end of sedation to extubation with no or minimal withdrawal symptoms | from end of sedation to extubation assessed up to 24 hrs

SECONDARY OUTCOMES:
To compare length of PICU stay in both groups | from Intubation to discharge assessed up to 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdullah Specialist Children Hospital (KASCH), Riyadh, Saudi Arabia